CLINICAL TRIAL: NCT06093412
Title: Application of Unilateral Epidural Anesthesia in Older Patients With Hip Fracture
Status: Completed | Type: Observational
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Peng Liu, Professor, Sichuan Provincial People's Hospital
Other Study IDs: h9mwa68d
Record Dates: First submitted 2023-09-29; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Spinal Anesthesia
Keywords: unilateral epidural anesthesia; combined lumbar and epidural anesthesia
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- unilateral epidural anesthesia (UEA) group: Patients were divided into two groups based on the type of anesthesia they received; a UEA group (n = 42) and a combined spinal epidural anesthesia (CSEA) group (n = 64).
  Interventions: Procedure: unilateral epidural anesthesia
- combined lumbar and epidural anesthesia (CSEA) group: Patients were divided into two groups based on the type of anesthesia they received; a UEA group (n = 42) and a combined spinal epidural anesthesia (CSEA) group (n = 64).
  Interventions: Procedure: combined lumbar and epidural anesthesia

INTERVENTIONS:
Procedure: unilateral epidural anesthesia — The patients received unilateral epidural anesthesia
  Groups: unilateral epidural anesthesia (UEA) group
Procedure: combined lumbar and epidural anesthesia — The patients received combined lumbar and epidural anesthesia
  Groups: combined lumbar and epidural anesthesia (CSEA) group

SUMMARY:
Because of population ageing, fragility fractures have become a huge burden on healthcare systems and wider society. Fractures result in a sharp drop in both short-term and long-term quality of life, they have a strong influence on activities of daily living and mobility, and they are associated with a significant increase in 1-year mortality (18%-36%). Surgery can benefit elderly patients with hip fractures to an extent, but it entails inevitable risks, particularly with respect to general anesthesia. In recent years unilateral spinal anesthesia has attracted attention due to the advantages of hemodynamic stability, reduced anesthetic dosage, and sufficient sensory block.

On the basis of a previous study, in the current study anesthetics were directly implanted into the unilateral epidural space in elderly patients with hip fractures prior to the completion of surgery. Data from 106 patients with old hip fractures who had undergone surgical treatment incorporating unilateral epidural anesthesia (UEA) or combined lumbar and epidural anesthesia were retrospectively analyzed in an attempt to provide a feasible solution for this kind of patients' anesthesia.

DETAILED DESCRIPTION:
Surgery can benefit elderly patients with hip fractures to an extent, but it entails inevitable risks, particularly with respect to general anesthesia. In recent years unilateral spinal anesthesia has attracted attention due to the advantages of hemodynamic stability, reduced anesthetic dosage, and sufficient sensory block. On the basis of a previous study, in the current study anesthetics were directly implanted into the unilateral epidural space in elderly patients with hip fractures prior to the completion of surgery.

ELIGIBILITY:
Inclusion Criteria:

had a fracture of a proximal femur were aged > 65 years the fracture occurred within 2 weeks of receiving treatment with comorbidities including pulmonary disease, arrhythmia, senile valve disease or lacunar infarction underwent intraspinal anesthesia during surgery

Exclusion Criteria:

had a secondary fracture after endoprosthetic reconstruction or intramedullary nail had a pathological fracture caused by tumor or tuberculosis condition was accompanied by lower limb nerve dysfunction had a cognitive or psychiatric disorder coagulation disorders hospitalization data were incomplete.

Ages: 66 Years to 94 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The totally 106 older patients (49 male, 57 female) aged 65-94 years with hip fractures who underwent surgery between January 2018 and June 2020 at the Orthopedic Department of our Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Hemodynamic change | Within 5 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 5 minutes after anesthesia
  Oxygen saturation
Hemodynamic change | Within 10 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 10 minutes after anesthesia
  Oxygen saturation
Hemodynamic change | Within 15 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 15 minutes after anesthesia
  Oxygen saturation
Hemodynamic change | Within 20 minutes after anesthesia
  Heart rate
Hemodynamic change | Within 20 minutes after anesthesia
  Oxygen saturation

SECONDARY OUTCOMES:
Dose of ephedrine use | During the surgery period
  Recoded dose of ephedrine use

OTHER OUTCOMES:
Duration of hospital stay | During the surgery period
  Recoded duration of hospital stay
Mortality | Perioperative period
  Mortality
Lower limb function | One year later
  Lower limb function (Harris score)

CONTACTS AND LOCATIONS:
Overall Officials: Overall Study Officials Zhao, M.D., Principal Investigator — Sichuan Provincial People's Hospital
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Prestmo A, Hagen G, Sletvold O, Helbostad JL, Thingstad P, Taraldsen K, Lydersen S, Halsteinli V, Saltnes T, Lamb SE, Johnsen LG, Saltvedt I. Comprehensive geriatric care for patients with hip fractures: a prospective, randomised, controlled trial. Lancet. 2015 Apr 25;385(9978):1623-33. doi: 10.1016/S0140-6736(14)62409-0. Epub 2015 Feb 5. PMID 25662415
- [Background] Cheng SY, Levy AR, Lefaivre KA, Guy P, Kuramoto L, Sobolev B. Geographic trends in incidence of hip fractures: a comprehensive literature review. Osteoporos Int. 2011 Oct;22(10):2575-86. doi: 10.1007/s00198-011-1596-z. Epub 2011 Apr 12. PMID 21484361
- [Background] Bentler SE, Liu L, Obrizan M, Cook EA, Wright KB, Geweke JF, Chrischilles EA, Pavlik CE, Wallace RB, Ohsfeldt RL, Jones MP, Rosenthal GE, Wolinsky FD. The aftermath of hip fracture: discharge placement, functional status change, and mortality. Am J Epidemiol. 2009 Nov 15;170(10):1290-9. doi: 10.1093/aje/kwp266. Epub 2009 Oct 4. PMID 19808632